CLINICAL TRIAL: NCT01678625
Title: Electromyographic Assessment of Onset and Recovery of Neuromuscular Blockade
Status: Terminated | Type: Observational
Why Stopped: Company making the device no longer in existence. Did not finish supplying data to research team
Sponsor: Endeavor Health (Other)
Collaborators: T4 Analytics (Industry)
Responsible Party: Principal Investigator, Glenn Murphy, Director, Clinical Research, Endeavor Health
Other Study IDs: EH12-158
Record Dates: First submitted 2012-08-28; First posted 2012-09-05 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Residual Neuromuscular Blockade
Keywords: Residual neuromuscular blockade; Train-of-four; Acceleromyography; Electromyography
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acceleromyography group: Train-of-four ratio calculation (TOF-Watch-SX-Bluestar enterprise)
  Interventions: Device: Train-of-four ratio calculation (T4-EMG)
- Electromyography group: Train-of-four ratio calculation (T4-EMG)
  Interventions: Device: Train-of-four ratio calculation (T4-EMG)

INTERVENTIONS:
Device: Train-of-four ratio calculation (T4-EMG) — TOF ratios will be compared between the EMG and AMG groups

SUMMARY:
Residual neuromuscular blockade (weakness) is a common occurrence in the postanesthesia care unit when muscle relaxant drugs have been used in the operating room. The only method of reliably detecting the presence of neuromuscular blockade is through the use of quantitative neuromuscular monitors. These devices measure and quantify the degree of muscle weakness and display the results on a screen. When using train-of-four (TOF) nerve stimulation, the ratio of the fourth muscle contraction (twitch) to the first twitch will be displayed; when this ratio is 90% (or 0.9) or greater, full recovery of muscle strength is present, and the endotracheal tube can be removed. At the present time, there is only one commercially-available quantitative monitor available in the United States -the TOF-Watch. It is not used by many clinicians because it requires experience to obtain accurate results, is expensive, and is subject to interference by factors in the operating room. The aim of this investigation is to examine a new quantitative monitor (the T4-EMG (EMG = electromyography) that may not be subject to the same limitations as the TOF-Watch AMG (AMG = acceleromyography). In order to study the accuracy of this new device, the T4-EMG will be compared to the current "clinical gold standard", the TOF-Watch.

DETAILED DESCRIPTION:
The aim of this investigation is to examine a new prototype of a quantitative monitoring instrument that will meet these requirements. Patients undergoing surgery under general anesthesia will be monitored with a new EMG device (T4-EMG) from induction of anesthesia until recovery of neuromuscular blockade. Continuous data will be recorded onto an interfaced computer from the T4-EMG monitor during this time period. At the same time, continuous neuromuscular data will be recorded onto the computer from an AMG device (TOF-Watch, the "established standard" for clinical use) which is attached to the same arm. The applicability (ease of use, equipment need, etc.), repeatability (precision or internal consistency), and performance (agreement with established standard, bias) of the T4-EMG compared to the AMG will be determined during onset and recovery of neuromuscular blockade.

44 patients presenting for elective surgical procedures with an expected duration greater than 60 minutes will be enrolled in this study. ASA I to III patients requiring neuromuscular blockade in the operating room will be eligible for enrollment. Anesthetic management will be standardized.

Upon arrival to the operating room, neuromuscular monitoring surface electrodes will be applied. All monitoring will be conducted while the patient is under general anesthesia for the surgical procedure. Surface electrodes (non-invasive EKG electrodes) will be placed on the cleansed skin over the ulnar nerve of the available arm near the wrist. The electrodes will be connected by leads to a peripheral nerve stimulator (TOF-Watch). When the nerve stimulator is activated, the response to stimulation will be measured simultaneously by the AMG (TOF-Watch-acceleration of contraction of the adductor pollicis-thumb) and the EMG (T4-EMG-electrical activity of the adductor pollicis-thumb) devices. Therefore, the TOF-Watch will serve as nerve stimulator for both study groups. The transducer of the AMG device will be placed on the thumb of the corresponding hand. A 75-150g preload (via the Hand adapter) will be applied as per standard recommendations. After induction of anesthesia, but before administration of rocuronium, calibration, supramaximal stimulation, and stable baseline will be achieved for the TOF-Watch as suggested by the GCRP guidelines.

The T4-EMG will be placed on the same arm as the AMG device, with sensing electrodes attached to the surface of the thenar eminence (base of the thumb). A second sensing lead, used to detect the delivery of an electrical stimulating pulse, will be placed over the stimulating leads of the AMG device. This sensing lead will only be used to trigger data acquisition in the T4-EMG, and has no direct connection to the patient, nor any electrical feedback connection that alters the function of the AMG. After a satisfactory level of stimulation and response has been obtained for the TOF-Watch, the T4-EMG device will be turned on, and the impedance of the thenar sensing leads will be measured. The trigger sense will be engaged, and further baseline stimuli will be delivered via the AMG (TOF-Watch). Data simultaneously collected from the thenar sensing leads will be inspected on the T4-EMG display, and fine adjustment of electrode positioning and stimulus intensity may be made to optimize the evoked myoelectric response from the patient. At the conclusion of the setup procedure, all settings of the AMG and the T4-EMG will be held constant for the remainder of the surgery.

After these baseline data are collected (average time 5 minutes), the neuromuscular blocking agent (NMBA) will be administered. Data relating to onset (a TOF ratio decreases from 1.0 to 0.3 or less on the AMG device display), maintenance (the TOF ratio is less than 0.3 and constant on the AMG device display), and reversal (an increase in the TOF ratio from 0.1 to 0.9 or above) will be recorded. Monitoring will continue until full recovery of neuromuscular function is noted (a TOF ratio of at least 0.9 or greater on the AMG device display). At this time, the anesthesia agents will be turned off and the patient awakened and extubated. Patients' trachea may extubated before achieving a TOF ratio of 0.9 if they awaken before this time, as per usual clinical routine determined by the clinician.

For the first 34 patients, the TOF-Watch is used as the nerve stimulator for both the AMG (TOF-Watch) and EMG (T4-EMG) groups. The ability of the T4-EMG device to sense/measure TOF ratios is the primary aim of the study (in comparison to the "clinical gold standard" TOF-Watch). However, the prototype T4-EMG (as well as the commercial device to be developed) will also contain a nerve stimulator (as do all qualitative and quantitative monitors). On a subset of patients monitored by the TOF-Watch (10 patients), the stand-alone T4-EMG device (single unit containing both the nerve stimulator and sensing/monitoring components) will be connected to the same arm and operated independently of the TOF-Watch. Its stimulating electrodes will be placed on the surface of the arm adjacent to the TOF-Watch electrodes; sensing leads will be placed on the thenar eminence as in the protocol described above. The T4-EMG will be set up independently of the TOF-Watch, with its own stimulator adjustment being made according to the same protocol as the TOF-Watch adjustment. The T4-EMG will be operated to stimulate and record at times selected by the anesthesiologist that do not conflict with operation of the TOF-Watch or interfere with other patient care activities. Evoked muscle response data will be displayed by the T4-EMG, but amplitude ratios will not be computed and it will not be used for direct patient care. The purpose is to demonstrate that the device elicits and records evoked muscle responses from surgical patients and to assess usability: this is in contrast to the main protocol where the T4-EMG is triggered by the TOF-Watch and where comparison of recorded responses is the goal.

The primary endpoint in the first 33 patients will be an analysis of the agreement between the AMG (clinical "gold standard") and EMG devices during neuromuscular recovery. Data will be compared between the two devices at AMG-derived TOF ratios values of 0.7, 0.8, 0.9, and 1.0 (if achieved) during recovery of neuromuscular function. Bias and limits of agreement will be calculated at each TOF value.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Status I to III patients requiring neuromuscular blockade in the operating room will be eligible for enrollment

Exclusion Criteria:

* 1) presence of an underlying neuromuscular disease; 2) use of drugs known to interfere with neuromuscular transmission (antiseizure medications, anticholinesterases, magnesium sulfate); 3) presence of renal or hepatic disease; or 4) procedures preventing access to at least one of the upper extremities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for elective surgical procedures under general anesthesia with an expected duration greater than 60 minutes will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Train-of-four (TOF)ratio | TOF ratios will be measured for the duration of the operation, approximately 3 hours
  Train-of-four ratios during recovery of neuromuscular blockade will be compared between the AMG and EMG devices (at a TOF ratio of 0.6, 0.7, 0.8, and 0.9.)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S. Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States